CLINICAL TRIAL: NCT05199441
Title: Efficacy and Tolerability of Galeo® in Patients With Postprandial Distress Syndrome Subtype in Functional Dyspepsia: a Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study
Brief Title: Efficacy of Galeo® in Patients With Postprandial Distress Syndrome Subtype in Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2021-034
Record Dates: First submitted 2021-12-17; First posted 2022-01-20 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dihydroxydibutylether group (Experimental): This group takes dihydroxydibutylether for 8 weeks.
  Interventions: Drug: Dihydroxydibutylether group
- Control group (Placebo Comparator): This group takes placebo for 8 weeks.
  Interventions: Drug: Control group placebo

INTERVENTIONS:
Drug: Dihydroxydibutylether group — This group takes 1.500 mg/day of dihydroxydibutylether for 8 weeks.
  Other Names: Galeo® group
  Arms: Dihydroxydibutylether group
Drug: Control group placebo — This group takes 1,500 mg/day of placebo for 8 weeks.
  Other Names: Placebo
  Arms: Control group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Galeo® on dyspepsia symptoms in patients with postprandial distress syndrome subtype in functional dyspepsia for 8 weeks.

DETAILED DESCRIPTION:
Galeo® already used an over-count drug for the improvement of dyspepsia symptoms. The investigators conduct a multi-center, double-blind, randomized, placebo-controlled, parallel-group study to investigate the effects of Galeo® on dyspepsia symptoms in patients with postprandial distress syndrome subtype in functional dyspepsia for 8 weeks; the safety of the compound is also evaluated. The Investigators examine gastrointestinal symptom score (GIS) score, the Korean version of Nepean dyspepsia index (K-NDI), and OV efficacy at baseline and after 8 weeks of intervention. A total of 226 subjects were administered either 1,500 mg of Galeo® or a placebo each day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* postprandial distress syndrome according to Rome III criteria
* Those who have at least 3 of the 10 symptoms of the GIS evaluation are moderate or more and have at least 1 of bloating, delayed digestion, belching, and nausea
* Those with no organic lesions on the upper gastrointestinal endoscopy within 3 months prior to screening

Exclusion Criteria:

* Those who have confirmed the following medical history or surgical history at the time of screening

  1. Surgery that may affect gastrointestinal motility (eg, laparoscopic or laparotomy of the gastrointestinal tract) (except for appendectomy and hysterectomy due to simple appendicitis)
  2. Diseases that can cause organic dyspepsia, such as irritable bowel syndrome, inflammatory bowel disease, gastroesophageal disease, and duodenal disease (gastric ulcer, esophagitis [from RE A], etc.) within 3 months before screening history of drug use
  3. Malignant tumors of the digestive system (except in cases where there is no history of recurrence within 5 years or cases where a cure has been obtained)
  4. Other malignant tumors other than the digestive system within 5 years (however, except for if there is no history of recurrence within 5 years or cured cases)
  5. History of organic neurological or psychiatric disorders (major depressive disorder or anxiety disorder, etc.), alcoholism, substance abuse, and drug dependence (except nicotine and caffeine)
* Those with the following diseases at the time of screening

  1. Organic causes of gastroparesis (diabetic gastroparesis, etc.)
  2. glaucoma
  3. urinary tract disease or prostate disease
  4. Biliary duct obstruction or biliary duct stones (eg, intrahepatic gallstones, extrahepatic gallstones)
  5. uncontrolled diabetes mellitus (glycated hemoglobin > 8.0%)
  6. Aspartate transaminase or alanine aminotransferase levels are more than 3 times the upper limit of normal, or total bilirubin levels are more than 3 times the upper limit of normal, or liver disease
  7. Serum creatinine level is 1.5 times or more of the upper limit of normal, or renal disease
  8. Other clinically significant diseases of the heart (blood pressure 160/100 mmHg or more), kidney, lung, blood, and endocrine system, and dysfunction that may affect efficacy and safety evaluation
* Those who have administered the following drugs that may affect efficacy evaluation within 2 weeks before screening

  1. emollient: artichoke extract, ursodeoxycholic acid, etc.
  2. prokinetics: metoclopramide, itopride, etc.
  3. inhibitors of gastric acid secretion: H2 receptor antagonist (proton pump inhibitor), gastric acid pump antagonist (acid pump antagonist)
  4. gastric mucosal protective agent, antacid, digestive agent
  5. fundus relaxants: sumatriptan, buspirone, etc.
  6. cholinergic, anticholinergic and antispasmodic
  7. psychotropic drugs: antipsychotic drugs, antidepressants, antimanic drugs, antianxiety drugs, hallucinogens, etc.
  8. Nonsteroidal anti-inflammatory drugs (intermittent administration up to 1 week 2 days and cyclooxygenase-2 selective inhibitors are acceptable)
  9. Antithrombotic agents (antiplatelet agents, anticoagulants)
  10. systemic glucocorticoids
  11. Erythromycin (However, in the case of eye drops, the administration is allowed) If the above drugs are administered, registration is possible after a wash-out period of at least 2 weeks, and drugs used for the purpose of pretreatment for upper gastrointestinal endoscopy (midazolam, propofol, simethicone), hyoscine butylbromide, cimetropium bromide, etc.) are allowed within 1 day.
* Those who received Helicobacter pylori eradication treatment within 2 weeks before screening
* Those who have administered or treated other clinical trial drugs or medical devices within 3 months prior to screening
* Pregnant or lactating women
* Women or men of childbearing potential who are unwilling to use an appropriate method of contraception* during this clinical trial

  *hormonal contraceptives, implantation of intrauterine devices or intrauterine systems, vasectomy, tubal ligation, double-blocking contraception (using a cervical cap or diaphragm and a male condom simultaneously), etc.
* If there are other diseases that may affect this clinical trial
* Persons with hypersensitivity or allergy to clinical investigational drugs and similar drugs or to soybean oil, soybean, peanut
* Persons judged unsuitable to participate in clinical trials by investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
gastrointestinal symptom total score at 4 weeks | 4 weeks
  Change in GIS total score at 4 weeks (Visit 4) compared to baseline (Visit 2). The minimum value was 0 and the maximum value was 40, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The Korean version of the Nepean Dyspepsia Index total score at 4 weeks | 4 weeks
  Change in the Korean version of the Nepean Dyspepsia Index total score at 4 weeks (Visit 4) compared to baseline (Visit 2). The minimum value was 0 and the maximum value was 195, and higher scores mean a worse outcome.
gastrointestinal symptom total score at 2 weeks | 2 weeks
  Change in GIS total score at 2 weeks (Visit 3) compared to baseline (Visit 2). The minimum value was 0 and the maximum value was 40, and higher scores mean a worse outcome.
Seven-point Likert scale for overall treatment efficacy at 4 weeks | 4 weeks
  Seven-point Likert scale for overall treatment efficacy evaluated by the subject at 4 weeks (Visit 4) after administration of the clinical trial drug. The minimum value was -3 and the maximum value was +3, and higher scores mean a better outcome.
each gastrointestinal symptom score at 2, 4 weeks | 2, 4 weeks
  Score change for each GIS symptom at 2 and 4 weeks (Visit 3, Visit 4) compared to the baseline (Visit 2). For each gastrointestinal symptom, the minimum value was 0 and the maximum value was 4, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No